CLINICAL TRIAL: NCT02200523
Title: Self Abrading Rapidly Applied (SARA) Electrode Phase II
Brief Title: Self Abrading Rapidly Applied Electrode Validation
Acronym: SARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Medical Devices Inc (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ns053116_SARA_electrode; R44NS053116 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-07-25 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: ELECTROENCEPHALOGRAPHIC VARIANT PATTERN 1 (Disorder)
Keywords: EEG; electrode

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SARA electrode (Experimental): new electrode
  Interventions: Device: SARA electrode
- Gold cup (Active Comparator): gold standard
  Interventions: Device: Gold cup

INTERVENTIONS:
Device: SARA electrode
  Arms: SARA electrode
Device: Gold cup
  Arms: Gold cup

SUMMARY:
The SARA (Self Abrading Rapidly Applied) electrode will speed EEG patient hookup by combining multiple steps that burden conventional EEG procedures into one. The investigators believe that the proposed system will reduce patient hookup time by more than 50% (from 40 to 20 minutes) with additional time savings on cleanup. Reducing the hookup time required for the EEG recording will make EEG more feasible in time critical situations and will improve patient care and service. The clinical testing in Phase II will investigate patient acceptance, clinician acceptance, time savings, and signal quality for 3 different environments: the large hospital institution, a small rural hospital setting and in an emergency department.

DETAILED DESCRIPTION:
The SARA (Self Abrading Rapidly Applied) electrode will speed EEG patient hookup by combining multiple steps that burden conventional EEG procedures into one. This proposed single-use electrode will consist of a Snap Top, Ag/AgCl Snap Conductor, Conductive Adhesive, and Abrader Tines in a custom molded housing and packed on a backing sheet. After removing the backing, the technician simply parts the hair with one hand and with the other hand rubs the electrode back and forth and then presses the electrode into position on the scalp. The proposed system combines the cumbersome and time-consuming skin preparation, electrode preparation and electrode fixation into one easy step. The investigators believe that the proposed system will reduce patient hookup time by more than 50% (from 40 to 20 minutes) with additional time savings on cleanup. Reducing the hookup time required for the EEG recording will make EEG more feasible in time critical situations and will improve patient care and service.

ELIGIBILITY:
Inclusion Criteria:

* adult and teenage

Exclusion Criteria:

* young children
* damaged scalp skin
* sensitive or allergic to electrode paste

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Weimer, Principal Investigator — Great Lakes NeuroTechnologies Inc.
Locations (1):
- MetroHealth Research Institute, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SARA Electrode: new electrode
  SARA electrode
- Gold Cup: gold standard
  Gold cup
Period: Overall Study
Arm/Group | SARA Electrode | Gold Cup
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SARA Electrode | Gold Cup | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: anonymous data did not include specific age information
Sex: Female, Male [Count of Participants; unit: Participants] — Population: anonymous data did not include gender information
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Signal Quality Comparison Between SARA Electrode and Gold Cup Electrode
Description: The time it takes in seconds to properly place the SARA electrodes and standard gold cup electrodes will be recorded and compared.
Time Frame: up to 1 hour
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SARA Electrode | Gold Cup
Number analyzed (Participants) | 20 | 20
seconds | 30 (10) | 45 (10)

ADVERSE EVENTS:
Time Frame: duration of the testing (<1 hour)
Description: ALL Adverse Events were monitored during the test by the clinician. Due to low risk of the procedure no subject was considered to be at risk for Mortality nor Serious Adverse Events but if one should occur during the test the clinician would observe and report.
Arm/Group | SARA Electrode | Gold Cup
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes